CLINICAL TRIAL: NCT06153706
Title: Evaluation of L-PRF as an Antibiotic Slow-release Biological Device in the Treatment of Moderate Periodontitis (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of L-PRF as an Antibiotic Slow-release Biological Device in the Treatment of Moderate Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yasmeen Khaled (Other)
Responsible Party: Sponsor-Investigator, Yasmeen Khaled, Periodontology Masters degree candidate, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #6/22
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-PFR loaded with medical grade metronidazole (Experimental)
  Interventions: Drug: Subgingival application of L-PRF loaded with metronidazole
- L-PFR (Active Comparator)
  Interventions: Other: Subgingival application of L-PRF

INTERVENTIONS:
Drug: Subgingival application of L-PRF loaded with metronidazole — After phase I therapy, L-PRF loaded medical grade metronidazole was applied sub gingivally into the pockets using blunt gauge needle and Perio-pack was placed (two applications with one week apart were applied subgingivally.
  Arms: L-PFR loaded with medical grade metronidazole
Other: Subgingival application of L-PRF — The L-PRF alone was applied subgingivally into the pockets and Perio-pack was placed (two applications with one week apart.
  Arms: L-PFR

SUMMARY:
This study aimed to evaluate the efficacy of leukocyte platelet-rich fibrin (L-PRF) as a local sustained released device for antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stage II periodontitis with probing depth and exhibiting bleeding on probing.
* Patients showing good oral hygiene.
* No history of periodontal therapy (surgical and non-surgical) for the past 6 months.

Exclusion Criteria:

* Patients with known systemic and debilitating diseases.
* Patients who had any previous adverse reactions to the products (or similar products) used in this study.
* Patients who have any autoimmune diseases.
* Patients who have any known disease that interfere with periodontal procedure.
* Smokers.
* Pregnancy and lactating women.
* Use of antibiotics during the last 6 months.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Plaque accumulation | up to 6 months
  This was assessed using O'Leary plaque index which is based on the visible continuous plaque along the gingival margin after staining. Four or six sites per tooth were examined, and the percentage of tooth surfaces exhibiting stained plaque was calculated. The score ranges from 0% (no plaque) to 100% (abundant plaque)
Gingival inflammation | up to 6 months
  This was assessed using modified gingival index which uses a visual scale to assess gingival health. It relies on a visual assessment of gingival changes to measure the severity of inflammation. Five categories, using a 0-4 scale, score the marginal and papillary gingival tissue based on color, texture, edema, and spontaneous bleeding. Using this index, 108 sites are scored per person (52 papillary and 56 marginal sites). Score 0 indicates normal gingival, score 1: mild inflammation with slight changes in color and texture, but not in all portions of gingival marginal or papillary, score 2: Mild inflammation with slight changes in color and texture in all portions of gingival marginal or papillary, score 3: Moderate bright surface inflammation, erythema, edema, and/or hypertrophy of gingival marginal or papillary, and score 4: Severe inflammation with erythema, edema, and/or marginal gingival hypertrophy of the unit or spontaneous bleeding, papillary, congestion, or ulceration
Bleeding on probing | up to 6 months
  This was assessed using bleeding index which assesses bleeding on probing. The number of sites where bleeding is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the bleeding index as a percentage. The score ranges from 0% (no bleeding) to 100% (bleeding in all sites)
Probing depth | up to 6 months
  The distance measured (mm) using a periodontal probe from the base of the pocket to the most apical point on the gingival margin. It dictates the patient's ability to maintain optimal plaque control. Probing depths in excess of 3mm are an indication for periodontal therapy.
Clinical attachment loss | up to 6 months
  It represents the extent of periodontal support that has been lost around a tooth and is measured with the periodontal probe as the distance (mm) from the cemento-enamel junction to the base of the pocket
Quantitative assessment of Porhyromonas gingivalis | up to 6 months
  Relative quantitation of Porhyromonas gingivalis counts was performed by Real Time PCR. Subgingival plaque samples were calculated, DNA was isolated and quantified for standardizing the polymerase chain reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmeen K Omar, BDS, Principal Investigator — Alexandria University; Mohy A El Rashidy, PhD, Study Director — Alexandria University; Ghada Bassiouny, PhD, Study Chair — Alexandria University; Aliaa G Aboulela, PhD, Study Chair — University of Alexandria
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Omar YK, Rashidy MAE, Ahmed GB, Aboulela AG. Evaluation of leukocyte-platelet rich fibrin as an antibiotic slow-release biological device in the treatment of moderate periodontitis: a randomized controlled clinical trial. BMC Oral Health. 2024 Dec 21;24(1):1530. doi: 10.1186/s12903-024-05254-x. PMID 39709402